CLINICAL TRIAL: NCT07198711
Title: Comparison of Ketamine Versus Saline During Sedation in Patients With Major Depressive Disorder: a Double-blind Trial
Brief Title: Induction of Dreaming With EEG and Anesthesia in Healthy Adults
Acronym: IDEA
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Tiny Blue Dot Foundation (Other)
Responsible Party: Principal Investigator, Boris D. Heifets, Associate Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 55215
Record Dates: First submitted 2025-09-14; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
Keywords: anesthesia; propofol; dreaming; consciousness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emergence-from-LOR Protocol (Experimental): Participants receive propofol titrated to loss of responsiveness (LOR) followed by maintenance and spontaneous emergence. This protocol is designed to elicit dream reports upon emergence (i.e., reports of subjective experiences occurring during the unresponsiveness period)
  Interventions: Drug: Propofol - Emergence-from-LOR Protocol
- No-LOR Light Sedation Protocol (Experimental): Participants receive propofol titrated stepwise to light sedation without LOR, maintaining responsiveness. This protocol is designed to elicit non-dream experiential reports while responsive (e.g., simple imagery, sounds, thoughts, bodily sensations, hypnagogic-like experiences).
  Interventions: Drug: Propofol - Light Sedation Protocol

INTERVENTIONS:
Drug: Propofol - Emergence-from-LOR Protocol — Intravenous propofol infusion that meets the criteria: (1) maintenance of spontaneous ventilation, (2) sedation level corresponding to a Patient State Index (PSI) no lower than 25; and (3) loss of responsiveness (LOR) defined by the Richmond Agitation Sedation Scale (RASS) = -5 [unarousable]. Anesthesia is then maintained at that level for 30 minutes, followed by spontaneous emergence.
  Arms: Emergence-from-LOR Protocol
Drug: Propofol - Light Sedation Protocol — Intravenous propofol infusion titrated stepwise to reach a state where participants are sedated but have behavioral responsiveness. Sedation is maintained at this level for 30 minutes.
  Arms: No-LOR Light Sedation Protocol

SUMMARY:
This open-label, randomized crossover study in healthy adults tests two propofol protocols to produce distinct experiential states. One induces brief loss of responsiveness with spontaneous emergence, intended to elicit dream reports; the other maintains light sedation without loss of responsiveness, intended to elicit non-dream experiences while participants remain responsive. The main goals are to (a) measure the protocol-concordant experiential report rate (how often each method produces its intended experience), (b) explore EEG correlates of these experiences in the two states, and (c) describe their phenomenology (what they are like). We will also examine short-term changes in well-being and sleep related to these experiences. Participants complete four sessions (two of each method) with EEG and routine monitoring, immediate post-session interviews, and brief questionnaires and daily sleep/dream logs before and after anesthesia sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 70 years of age, inclusive, at screen.
2. Able to read, understand, and provide written, dated informed consent prior to screening. Participants will be deemed likely to comply with study protocol and communicate with study personnel about adverse events and other clinically important information.
3. In sufficiently good health to proceed with a low risk elective procedure, characterized using the American Society of Anesthesiologists (ASA) physical status classification system as Class 1 or 2.
4. If female, a status of non-childbearing potential or use of an acceptable form of birth control
5. Body mass index between 17-35 kg/m2.

Exclusion Criteria:

1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
2. Female that is pregnant or breastfeeding.
3. Female with a positive pregnancy test at screening or baseline.
4. Current diagnosis of a Substance Use Disorder (SUD; Abuse or Dependence, as defined by DSM-V) rated "moderate" or "severe", or Alcohol Use Disorder rated "moderate" or "severe". The following categories of SUD will NOT be excluded: nicotine dependence; alcohol or substance use disorder rated "mild"; alcohol or substance use disorder of any severity in remission, either early (3-12 months) or sustained (>12 months) time frames.
5. Current diagnosis of Axis I disorders other than Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, Specific Phobia, or Bipolar II Disorder
6. History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms
7. History of anorexia nervosa, bulimia nervosa, or eating disorder not otherwise specified, within five years of screening.
8. In the judgment of the investigator, the subject is at significant risk for suicidal behavior during the course of his/her participation in the study.
9. A neurological disorder including:

   1. Has dementia, delirium, amnestic, or any other cognitive disorder.
   2. Lifetime history of surgical procedures involving the brain or meninges,
   3. encephalitis, meningitis, degenerative central nervous system disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation
   4. any other disease/procedure/accident/intervention associated with significant injury to or malfunction of the central nervous system (CNS),
   5. history of significant head trauma within the past two years.
10. A cardiovascular disorder including:

    1. uncontrolled hypertension
    2. Congestive heart failure NYHA Criteria >Stage 2
    3. Atrial fibrillation or resting heart rate <50 or >105 beats per minute at screening or randomization
    4. Any conduction abnormalities including AV nodal block of any type or intraventricular conduction delay.
    5. QTcF (Fridericia-corrected) >= 450 msec at screening or randomization
    6. any cardiovascular disorder that would merit categorization of patient as ASA Class 3 or higher
11. A pulmonary/respiratory disorder including:

    1. diagnosed Obstructive Sleep Apnea or STOPBANG score of 3 or higher
    2. History of difficult airway in surgical setting
    3. any pulmonary / respiratory disorder that would merit categorization of patient as ASA Class 3 or higher
12. Clinically significant liver disease, determined by LFTs within the past 6 months.
13. Clinically significant kidney disease determined by creatinine / GFR within the past 6 months.
14. Symptomatic gastroesophageal reflux disease, hiatal hernia, or other gastrointestinal disorder placing patient at risk for aspiration or that would merit categorization of patient as ASA Class 3 or higher
15. Any endocrine disorder including:

    1. uncontrolled diabetes, type 1 or 2
    2. History of hypothyroidism and has been on a stable dosage of thyroid replacement medication for less than six months prior to screening. (Subjects on a stable dosage of thyroid replacement medication for at least six months or more prior to screening are eligible for enrollment.)
    3. History of hyperthyroidism which was treated (medically or surgically) less than six months prior to screening.
    4. Other endocrine disorder that would merit categorization of patient as ASA Class 3 or higher
16. Patients taking any of the following daily medications:

    1. opioids including buprenorphine and methadone
    2. naltrexone or other opioid antagonist
    3. clonidine
17. Any other clinically significant abnormal laboratory result at the time of the screening exam.
18. Has a clinically significant abnormality on the screening physical examination that might affect safety, study participation or confound interpretation of study results, including any condition that would merit categorization of patient as ASA Class 3 or higher.
19. Participation in any clinical trial with an investigational drug or device that conflicts with this trial, within the past month or concurrent to study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Protocol-concordant experiential report | Assessed within 5 minutes of return of responsiveness (LOR protocol) or within 5 minutes of session end (light-sedation protocol).
  Presence vs absence of an experiential report elicited via a structured interview (modified Brice). "Protocol-concordant" is defined as:
  LOR protocol-success = any dream report upon emergence; Light-sedation (no-LOR) protocol-success = any experiential report that is not a dream (e.g., imagery, sounds, thoughts, bodily sensations, hypnagogic-like experiences) while the participant remained behaviorally responsive.

SECONDARY OUTCOMES:
EEG correlates of protocol-concordant experiential outcome | Matched-duration EEG windows during the 30-minute maintenance period: pre-emergence window prior to return of responsiveness in the LOR protocol, and a time-matched window during maintenance in the no-LOR protocol.
  EEG correlates of the two protocols/states, examining spectral band powers, band ratios, and other features during the matched windows and their association with protocol-concordant experiential outcomes.
Phenomenology of anesthesia experiences (analysis of narrative reports) | Interview immediately post-session
  Transcriptions of audio-interviews and analysis of these using (i) codebook-based content analysis, (ii) phenomenological thematic/structural coding, and (iii) NLP-derived text features.
Phenomenology of anesthesia experiences (self-ratings) | Interview immediately post-session
  Participants' own ratings of their anesthesia experiences: complexity, vividness, affect (valence/intensity), meaningfulness, dynamism/movement, bizarreness, perceived duration, the degree of mystical experiences (Mystical Experience Questionnaire; Barrett et al., 2015) and challenging experiences (Challenging Experience Questionnaire; Strickland et al., 2024).
Dream vs dream-like experiences (within-anesthesia) - phenomenological differences | Interview immediately post-session
  Comparison of phenomenology between anesthesia dreams (LOR protocol) and dream-like experiences (light sedation no-LOR protocol) based on the analysis of narrative reports and self-ratings of the experiences
Home dreams vs anesthesia dreams - phenomenological differences | Home dream logs (2 weeks pre-session and 2 weeks post-session) vs anesthesia interview (immediate post-session).
  Differences in phenomenology of home dreams vs anesthesia dreams based on the analysis of narrative reports and self-ratings of these experiences
Safety outcomes | From pre-anesthesia baseline to post-anesthesia discharge
  Incidence of adverse events during anesthesia or recovery (e.g., PONV; hypoxemia; hypotension; airway intervention) and any serious adverse events per FDA criteria.
Changes in daily mood | Baseline (2-week pre-session average) to follow-up (2-week post-session average)
  As measured with the following mood scales: PANAS (Watson et al., 1988) and items from the 12-point Affect Circumplex (Yik et al., 2011)
Change in well-being: life satisfaction | Baseline (2-weeks pre-anesthesia) to follow-up (2-weeks post-anesthesia)
  As measured with The Satisfaction With Life Scale (Diener et al., 1985)
Change in well-being: peace of mind | Baseline (2-weeks pre-anesthesia) to follow-up (2-weeks post-anesthesia)
  As measured with The Peace of Mind Scale (Lee et al., 2013)
Change in sleep quality | Baseline (2-week pre-session) to follow-up (2-week post-session)
  Change in sleep quality as measured using the Pittsburgh Sleep Quality Inventory (PSQI; Buysse et al., 1989) and daily sleep and dream diaries
Change in dream outcomes | Baseline (2-week pre-session) to follow-up (2-week post-session).
  Change in dream recall frequency, occurrence of nightmares, nightmare distress as measured using the Mannheim Dream Questionnaire (MADRE; Schredl et al., 2014) and daily dream diaries
Change in well-being: harmony in life | Baseline (2-weeks pre-anesthesia) to follow-up (2-weeks post-anesthesia)
  As measured with the Harmony in Life Scale (Kjell et al., 2016)
Change in well-being: psychological (eudaimonic) well-being | Baseline (2-weeks pre-anesthesia) to follow-up (2-weeks post-anesthesia)
  As measured with the Psychological Well-Being Scale (Ryff, 1989)
Change in alexithymia score | Baseline (2-weeks pre-anesthesia) to follow-up (2-weeks post-anesthesia)
  As measured with the Perth Alexithymia Questionnaire Short Form (Preece et al., 2023)
Change in emotion regulation | Baseline (2-weeks pre-anesthesia) to follow-up (2-weeks post-anesthesia)
  As measured with the Emotion Regulation Questionnaire (Gross & John, 2003) and the Perth Emotion Regulation Competency Index (Preece et al., 2018)
Change in symptoms of depression | Baseline (2-weeks pre-anesthesia) to follow-up (2-weeks post-anesthesia)
  As measured with the depression module of the Patient Health Questionnaire (PHQ9; Spitzer et al., 1999)
Change in symptoms of anxiety | Baseline (2-weeks pre-anesthesia) to follow-up (2-weeks post-anesthesia)
  As measured with the The Generalized Anxiety Disorder Scale (GAD-9; Spitzer et al., 2006)
Change in perceived loneliness | Baseline (2-weeks pre-anesthesia) to follow-up (2-weeks post-anesthesia)
  As measured the 3-item UCLA Loneliness Scale (Hughes et al., 2004)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Boris D Heifets, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Identifiers might be removed from identifiable private information and/or identifiable specimens and, after such removal, the information and/or specimens could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from the participant.
  The results of this research study may be presented at scientific or medical meetings or published in scientific journals without disclosing the identify of the participants (unless there is a separate consent from participants to reveal their identity).
Supporting Information: Study Protocol
Time Frame: After the completion of the study and upon publishing the results

REFERENCES:
- [Background] Chow HS, Hack LM, Kawai M, Heifets BD. Anesthetic-Induced Intraoperative Dream Associated With Remission of a Psychiatric Disorder: A Case Report. A A Pract. 2022 Aug 10;16(8):e01613. doi: 10.1213/XAA.0000000000001613. eCollection 2022 Aug 1. PMID 35952341
- [Background] Hack LM, Sikka P, Zhou K, Kawai M, Chow HS, Heifets B. Reduction in Trauma-Related Symptoms After Anesthetic-Induced Intra-Operative Dreaming. Am J Psychiatry. 2024 Jun 1;181(6):563-564. doi: 10.1176/appi.ajp.20230698. Epub 2024 Mar 13. No abstract available. PMID 38476046